CLINICAL TRIAL: NCT05717920
Title: The ADRO Trial: An Adaptive, 2-Part, Phase 2 Clinical Trial Investigating the Safety and Efficacy of ADX-629 in Adults With Atopic Dermatitis
Brief Title: A Clinical Trial in Subjects With Atopic Dermatitis (Part 1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADX-629-ATD-001
Record Dates: First submitted 2023-01-25; First posted 2023-02-08 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Atopic Dermatitis
Keywords: eczema; atopic; adaptive; Aldeyra; ADX-629; Reactive aldehyde species (RASP)
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — ADX-629

STUDY DESIGN:
Masking Description: Part 1 is an open-label trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADX-629 (Experimental)
  Interventions: Drug: ADX-629 (Open-label)

INTERVENTIONS:
Drug: ADX-629 (Open-label) — ADX-629 (250 mg) administered twice daily for 90 days

SUMMARY:
A Phase 2, multicenter, adaptive 2-part clinical trial designed to evaluate the safety and efficacy of ADX-629 alone and in combination with standard-of-care in adults with atopic dermatitis.

DETAILED DESCRIPTION:
The trial is divided into 2 parts; the first part of the trial (Part 1) is open label, and the second part (Part 2) is randomized, double-blind, and placebo controlled.

In Part 1, approximately 10 subjects will receive open-label ADX-629 twice daily for 90 days.

In Part 2, approximately 40 subjects will be randomized to receive either ADX-629 or matching placebo twice daily for 90 days.

Patients who are interested in participating will be provided detailed information about the study including description of study assessments/procedures, possible side-effects, alternative treatments, and potential benefits.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* History of atopic dermatitis, according to American Academy of Dermatology criteria, that has been present for at least 6 months
* Mild, moderate, or severe atopic dermatitis, defined as an IGA score of ≥2 at Baseline
* Not pregnant, breastfeeding, or lactating and agree to use a highly effective method of acceptable contraceptive for the trial duration, if applicable

Exclusion Criteria:

* Presence of clinically significant kidney disease or an estimated gloverular filtration rate (eGFR) of less than or equal to 45 milliliters/min/1.73 m2 during screening
* History of any unstable chronic diseases/conditions, clinically significant abnormalities, or findings, that in the opinion of the Investigator, could compromise subject safety or affect the conduct of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Adverse Event (AE) Query | From Day 1 to Day 90
  Incidence and severity of AEs

SECONDARY OUTCOMES:
Investigator Global Assessment (IGA) Score | From Day 1 to Day 90
  Change from Baseline in IGA Score

CONTACTS AND LOCATIONS:
Locations (1):
- Bexley Dermatology Research, Bexley, Ohio, United States

IPD SHARING:
Plan to Share IPD: No